CLINICAL TRIAL: NCT06229054
Title: Efficacy of Dexmedetomidine as an Adjuvant in Obturator Nerve Block for Postoperative Pain in Patients Undergoing Transurethral Surgeries Under Spinal Anesthesia : A Randomized Controlled Study
Brief Title: Dexmedetomidine in Obturator Nerve Block as an Analgesic in Transurethral Surgeries
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Karim Hussein, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DEX in obturator nerve block
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Dexmedetomidine
Keywords: obturator nerve block; Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group Dexmedetomidine (Experimental): : Patients in this group will receive regional anesthesia and obturator nerve block bilaterally (10 ml 2% preservative-free lignocaine along with 5 ml 0.5% preservative-free bupivacaine) and dexmedetomidine 100 mcg/mL (2µg/kg).
  Interventions: Drug: Dexmedetomidine; Drug: Bupivacaine Hydrochloride
- group Bupivacaine (Other): :Patients in this group will receive regional anesthesia and bilateral obturator nerve block only (10 ml 2% preservative-free lignocaine along with 5 ml 0.5% preservative-free bupivacaine).
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine (DEX), an α2-agonist with more promising pharmacokinetic and pharmacodynamic characteristics than clonidine has been proved to have a positive effect on postoperative pain intensity and to reduce opioid consumption
  Other Names: DEX
  Arms: group Dexmedetomidine
Drug: Bupivacaine Hydrochloride — local anesthesic which works through blocking sodium channels
  Other Names: marcaine

SUMMARY:
in our study, we will investigate the impact of adding dexmedetomidine to bupivacaine for the potency of the obturator nerve block and prevention of the postoperative pain associated with transurethral surgery in comparison of obturator nerve block with bupivacaine alone

DETAILED DESCRIPTION:
* After history taking and examination of the labs and airway of the patient , An intravenous catheter will be secured in the dorsum of the hand of non dominant hand and patients will be monitored for heart rate, noninvasive blood pressure, and oxygen saturation.
* All patients after aseptic preparation will receive subarachnoid block in lumber 3-4 or 4-5 space in sitting position.
* About 3 ml (15mg) of heavy 0.5% bupivacaine will be injected into subarachnoid space.
* After the completion of the block, patients will be laid in the supine position and subsequently waited for 5 min for fixation of drug and assessed for sensorimotor block.
* Further procedure will be performed as per the group allocation.
* ONB will be performed by classic technique 1.5cm lateral and 1.5cm caudal to the pubic tuberacle . after contact with the pubic ramus is made , the needle is redirected laterally to a point 2-3 cm deeper than the pubic ramus.(15)
* A waiting period 20 min will be allowed for the full effect of the block and then resection will be allowed to perform
* Hemodynamics (heart rate, mean arterial blood pressure) will be recorded intraoperatively and postoperative at 0, 2 and 6 hours .
* VAS score at 0,2 and 6 hours post-operatively will be assessed.
* Time to first call for analgesic requirements (duration of analgesia) will be measured.
* Total postoperative analgesic consumption in the first 24 hours post-operative will be measured.
* Incidence of complications such as nerve injury, hematoma formation, local anesthetic toxicity, intravascular injection, bleeding and bladder perforation will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be adults (above 18 years) scheduled to undergo transurethral surgery under regional anesthesia.
* ASA1, ASA2

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical class 3,4, severe cardiac comorbidity (impaired contractility with ejection fraction less than 50%, heart block, significant arrhythmias, tight valvular lesions), allergy to any study's drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Severity of pain measured by visual analog scale (VAS) score. postoperative pain after transurethral surgeries | 24 hours postoperatively
  the VAS score consists of 10cm line where 0 represents NO PAIN and 10 represents SEVEREST FORM OF PAIN

SECONDARY OUTCOMES:
• Perioperative analgesic consumption, which will be calculated as the total amount of opioids administered in the postoperative periods. | 24 hours postoperative
  to detect incidence of pain postoperative
• Incidence of adverse effects as bleeding and bladder perforation. | 24 hours postoperative
  to detect any complications occured during the surgery
• Incidence of adductor jerk reflex | intraoperative
  to detect incidience of jerk reflex during the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine-Cairo Univeristy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Badrinath R., Konety MD, MBA, Peter R., Carroll MD: Urothelial carcinoma in Smith's General Urology, edited by Emil A. Tanagho, Jack W., and MC Ninch (Eds.), 17th edition, MC Graw Hil, 2008.
- [Background] Peter T. Nich, MD; Fray F. Marshall, MD Surgery for bladder cancer. Walsh, Patrick C., Retik, Alan B., E. Darracott Vaughan, and Alan J. Wein [Eds]: Campbell's Urology, 9th ed. Philadelphia: Saunders, 2007. 2478
- [Background] Erbay G, Akyol F, Karabakan M, Celebi B, Keskin E, Hirik E. Effect of obturator nerve block during transurethral resection of lateral bladder wall tumors on the presence of detrusor muscle in tumor specimens and recurrence of the disease. Kaohsiung J Med Sci. 2017 Feb;33(2):86-90. doi: 10.1016/j.kjms.2016.11.006. Epub 2016 Dec 30. PMID 28137416
- [Background] Bilotta F, Pugliese F. The evolving clinical use of dexmedetomidine. Lancet. 2020 Jul 18;396(10245):145-147. doi: 10.1016/S0140-6736(20)30902-8. No abstract available. PMID 32682463
- [Background] Abdulatif M, Mukhtar A, Obayah G. Pitfalls in reporting sample size calculation in randomized controlled trials published in leading anaesthesia journals: a systematic review. Br J Anaesth. 2015 Nov;115(5):699-707. doi: 10.1093/bja/aev166. Epub 2015 Jun 3. PMID 26041717